CLINICAL TRIAL: NCT07054463
Title: Fu's Subcutaneous Needling-assisted Conservative Treatment for Distal Radius Fracture Healing: Protocol for a Randomized Controlled Trial
Brief Title: Clinical Study on the Healing of Distal Radius Fractures With Conservative Treatment Assisted by Fu's Subcutaneous Needling
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Cheng Chen, Principal Investigator, Guangzhou University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YF2025-126-01
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-04

CONDITIONS: Distal Radius Fractures
Keywords: Fu's subcutaneous needle therapy; distal radius fractures; conservative treatment
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSN Therapy Combined with Rehabilitation Training Group (Experimental): Patients randomized to the FSN group will receive additional FSN therapy to the immobilized region alongside standard rehabilitation. Prior to treatment, blinding will be ensured through the use of eye masks. The treatment protocol will consist of 12 sessions over 8 weeks: three sessions in the first week (administered every other day), two weekly sessions during weeks 2-3, and one weekly session during weeks 4-8.
  Interventions: Other: FSN Therapy Combined with Rehabilitation Training
- Sham FSN Combined with Rehabilitation Training Group (Sham Comparator): Patients randomized to this group will undergo the sham intervention in the same predetermined anatomical region. Prior to the procedure, eye masks will be applied to ensure blinding. The Sham FSN device, featuring a blunt tip, will generate a pricking sensation upon spring-loaded actuator deployment without actual skin penetration, maintaining parallel alignment to the epidermal surface. The treatment protocol will consist of 12 sessions over 8 weeks: three sessions in the first week (administered every other day), two weekly sessions during weeks 2-3, and one weekly session during weeks 4-8.
  Interventions: Other: Sham FSN Therapy Combined with Rehabilitation Training

INTERVENTIONS:
Other: FSN Therapy Combined with Rehabilitation Training — Prior to treatment, blinding will be ensured through the use of eye masks. Based on the "affected muscle theory," all forearm muscles within the splint-immobilized area will be considered as an affected muscle group and further subdivided into "flexor" and "extensor" subgroups according to functional anatomy.
  Two needle insertion points will be selected approximately 5 cm distal to the cubital crease, corresponding to the flexor and extensor muscle groups.
  Following standard disinfection of the insertion device and sites, a disposable FSN needle will be inserted subcutaneously into the superficial fascial layer, with the needle tip directed toward the affected muscle group. The needle core will then be retracted into the soft tube, ensuring no tip exposure, and the tube base will be secured within the handle slot. A 30° fan-shaped sweeping motion will be performed bilaterally at a frequency of 100 sweeps/min for 2 minutes.
  Arms: FSN Therapy Combined with Rehabilitation Training Group
Other: Sham FSN Therapy Combined with Rehabilitation Training — Patients randomized to this group will undergo the sham intervention in the same predetermined anatomical region. Prior to the procedure, eye masks will be applied to ensure blinding. The Sham FSN device, featuring a blunt tip, will generate a pricking sensation upon spring-loaded actuator deployment without actual skin penetration, maintaining parallel alignment to the epidermal surface.
  Following standard aseptic preparation, the acupuncturist will stabilize the needle body with the non-dominant hand while simulating insertion motions with the dominant hand, replicating the authentic FSN technique by retracting the stylet to the locking groove. The practitioner will then perform sweeping manipulations (ensuring continuous dermal contact during the procedure). Both the operational protocol and treatment course will be identical to those of the genuine FSN intervention group.
  Arms: Sham FSN Combined with Rehabilitation Training Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Fu's subcutaneous needling (FSN) therapy combined with rehabilitation exercises in promoting fracture healing after conservative treatment of distal radius fractures (DRFs) in adult patients (aged 18-85 years) with acute DRFs. The main questions it aims to answer are:

* Does FSN therapy accelerate radiographic union compared to Sham FSN therapy?
* Does FSN therapy improve functional outcomes (e.g., pain, swelling, joint mobility) and anatomical stability (e.g., volar tilt, radial height) in DRF patients?

Researchers will compare the FSN therapy plus rehabilitation training group to the Sham FSN therapy plus rehabilitation training group to see if FSN provides superior clinical benefits in fracture healing and functional recovery.

Participants will:

1. Receive either FSN or Sham FSN therapy (12 sessions over 8 weeks) alongside standardized rehabilitation exercises.
2. Undergo periodic assessments (weeks 2, 4, 6, 8, 10, and 12) for radiographic union, pain (VAS), swelling, wrist mobility, and functional status (DASH questionnaire).
3. Follow a phased rehabilitation protocol, including finger/shoulder exercises (weeks 1-3), gentle wrist movements (weeks 4-5), and resistance training (week 6 onward).

ELIGIBILITY:
Inclusion Criteria:

Participants meeting the diagnostic criteria for distal radius fractures as outlined in both the Evidence-Based Guidelines for Diagnosis and Treatment of Adult Distal Radius Fractures (2024) (10) and the clinical practice guidelines (CPG) jointly issued by the American Academy of Orthopaedic Surgeons (AAOS) and the American Society for Surgery of the Hand (ASSH) (11), while also satisfying the following conditions, will be eligible for enrollment:

1. Within 1 week post closed reduction and small splint immobilization treatment.
2. Aged between 18 and 85 years (inclusive).
3. Fracture caused by trauma.
4. Acute fracture (≤2 weeks) or first-time fracture.
5. No prior history of receiving Fu's subcutaneous needling therapy.
6. Signed informed consent form obtained.

Exclusion Criteria:

1. Pathological, open, or nonacute fractures (>2 weeks since injury).
2. Patients with thrombocytopenia, bleeding tendency, or coagulation disorders (INR >1.5 or platelet count <50×10⁹/L).
3. Cognitive impairment or psychiatric disorders affecting treatment compliance and follow-up.
4. Local skin lesions, pregnancy, or lactation.
5. History of syncope during Fu's subcutaneous needling therapy or intolerance to the procedure.
6. Participation in other interventional clinical trials within the past 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
the modified Radiographic Union Scale for Tibial Fractures (RUST) | From enrollment to the end of treatment at 8 weeks
  The modified RUST (Radiographic Union Scale for Tibial fractures) scoring system will be utilized to evaluate each of the four cortices on both anteroposterior and lateral wrist radiographs, assigning scores of 1 (no callus), 2 (presence of callus), 3 (bridging callus), or 4 (fracture remodeled and no longer visible). The sum of the four cortical scores yields a total ranging from 4 to 16 points, with a score of 13 points indicating fracture union. Assessments will be conducted at baseline, as well as at 2, 4, 6, and 8 weeks post-treatment. Time to osseous consolidation will be expressed as the median duration with the corresponding interquartile range (IQR).

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | From enrollment to the end of treatment at 8 weeks
  Scored from 0 to 10, with higher scores indicating more severe pain.
Swelling Severity Scale | From enrollment to the end of treatment at 8 weeks
  Graded as 0 (no swelling), 1 (mild swelling), 2 (moderate swelling), or 3 (severe swelling).
Wrist Joint Range of Motion (ROM) | From enrollment to the end of treatment at 8 weeks
  Measured using a goniometer for dorsiflexion, palmar flexion, radial deviation, and ulnar deviation.
Disabilities of the Arm, Shoulder and Hand (DASH) | From enrollment to the end of treatment at 8 weeks
  The DASH questionnaire is a tool used to assess upper limb functional status, symptom severity, and disability levels. It consists of 30 items evaluating difficulties in performing physical activities due to upper limb problems during the past week, including the severity of activity-related pain, symptoms such as pain, numbness, stiffness, and weakness, as well as the impact on work, daily activities, sleep, and psychological state. The DASH score ranges from 0 to 100, with higher scores indicating more severe disability.
Radial height | From enrollment to the end of treatment at 8 weeks
  On posteroanterior (PA) wrist radiographs, the distance between the tip of the radial styloid process and a line connecting the dorsal and volar edges of the lunate fossa, perpendicular to the longitudinal axis of the radial shaft.
Ulnar Variance | From enrollment to the end of treatment at 8 weeks
  On posteroanterior (PA) wrist radiographs, the distance between two lines perpendicular to the longitudinal axis of the radius: one at the level of the distal radial articular surface and the other at the most distal point of the ulnar head.
Radial Inclination (Ulnar Deviation Angle) | From enrollment to the end of treatment at 8 weeks
  On posteroanterior (PA) wrist radiographs, the angle between a line connecting the tip of the radial styloid process and the midpoint of the dorsal and volar edges of the lunate fossa, and a line perpendicular to the longitudinal axis of the radial shaft.
Volar Tilt (Palmar Inclination Angle) | From enrollment to the end of treatment at 8 weeks
  On lateral wrist radiographs, the angle between a line connecting the most distal points of the volar and dorsal articular surfaces and a line perpendicular to the longitudinal axis of the distal radius.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Sun, Principal Investigator — Guangzhou University of Chinese Medicine - Department of Acupuncture and Rehabilitation Clinical Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR